CLINICAL TRIAL: NCT06526702
Title: Intradialytic Kinetics of Cardiac Biomarkers During Hemodialysis and Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Hundborg Liboriussen, Principal Investigator, Medical Doctor, and PhD student at the Department of Nephrology, Aalborg University Hospital, Denmark, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: F2024-045 and N-20240016
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Renal Dialysis; Hemodiafiltration; Hemodialysis; Peritoneal Dialysis; Renal Replacement Therapy; Troponin; Natriuretic Peptide, Brain; Secretoneurin; Biomarkers; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, crossover study with 24 participants. The study will investigate the effect of high-flux hemodialysis (using the FX CorDiax 100 dialyzer) and post-dilution HDF (using the FX CorDiax 1000 dialyzer) on the intradialytic kinetics of selected cardiac biomarkers. The study will not be blinded, but the order of the interventions will be randomized. The two dialysis sessions will be conducted on the same weekday. Between the two interventions, the patient will have a wash-out period of 1-3 weeks with standard dialysis treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-flux hemodialysis then post-dilution hemodiafiltration (Experimental): Participants will first receive high-flux hemodialysis. Following a washout period of 1-3 weeks, they will receive post-dilution hemodiafiltration.
  Interventions: Device: High-flux hemodialysis; Device: Post-dilution hemodiafiltration
- Post-dilution hemodiafiltration then high-flux hemodialysis (Experimental): Participants will first receive post-dilution hemodiafiltration. Following a washout period of 1-3 weeks, they will receive high-flux hemodialysis.
  Interventions: Device: High-flux hemodialysis; Device: Post-dilution hemodiafiltration

INTERVENTIONS:
Device: High-flux hemodialysis — FX CorDiax 100 dialyzer
Device: Post-dilution hemodiafiltration — FX CorDiax 1000 dialyzer

SUMMARY:
This randomized, crossover study aims to investigate the intradialytic kinetics of selected cardiac biomarkers in patients with end-stage renal disease treated with dialysis. The cardiac biomarkers of interest include high-sensitivity cardiac troponin I, high-sensitivity cardiac troponin T, brain natriuretic peptide, and a novel cardiac biomarker named secretoneurin.

In 24 patients treated with maintenance hemodialysis, the study will compare high-flux hemodialysis (HD) with post-dilution hemodiafiltration (HDF) to investigate:

* Baseline concentrations and week-to-week plasma variations of the cardiac biomarkers.
* Changes in the plasma concentrations of the cardiac biomarkers during high-flux HD and post-dilution HDF.
* Dialyzer clearance of the cardiac biomarkers in high-flux HD and post-dilution HDF.
* Adherence of the cardiac biomarkers to the dialyzer membrane.
* Concentrations of the cardiac biomarkers 30 minutes post-dialysis to investigate a potential rebound effect.

Additionally, a sub-study of 24 patients treated with peritoneal dialysis will investigate the baseline concentrations and week-to-week plasma variations of the same cardiac biomarkers.

DETAILED DESCRIPTION:
Patients treated with maintenance hemodialysis:

Single-center, randomized, crossover study with 24 participants. The study will investigate the effect of high-flux HD (using the FX CorDiax 100 dialyzer) and post-dilution HDF (using the FX CorDiax 1000 dialyzer) on the intradialytic kinetics of selected cardiac biomarkers. The study will not be blinded, but the order of the interventions will be randomized. The two dialysis sessions will be conducted on the same weekday. Between the two interventions, the patient will have a wash-out period of 1-3 weeks with standard dialysis treatment.

On both trial days, the following dialysis settings will be the same for each individual patient:

* The dialysis sessions will last 4 hours.
* The same dialysis machine will be used, either the Fresenius Medical Care 5008 or 6008 CAREsystem machine.
* Same vascular access will be used.
* The composition of electrolytes in the dialysate will be the same.
* Blood flow rate will be >300 mL per minute and consistent.
* Dialysate flow rate will be 500 mL per minute.
* Ultrafiltration rate will be constant aiming at dry weight.
* Routine anticoagulation protocol will be unchanged, but consistent on both trial days.
* Routine dialysate temperature will be unchanged, but consistent on both trial days.

On both trial days, different baseline characteristics will be gathered, including demographic data, clinical data, dialysis characteristics, and routine blood samples. Blood samples, for the analysis of the selected cardiac biomarkers, will be collected:

* Before the dialysis session is started (baseline).
* After 10, 30, 60, 120, 180, and 240 minutes of dialysis. All samples will be collected from the blood dialyzer inlet; however, halfway into the dialysis session (after 120 minutes), samples will also be collected from the blood dialyzer outlet and from the dialysate.
* 30 minutes after dialysis cessation. However, if the patient will not stay 30 minutes, the post-dialysis sample will be gathered after 5 minutes.

Sub-study of patients treated with peritoneal dialysis:

In a sub-study, 24 patients treated with peritoneal dialysis, will be included for one or two venous blood samples (with a minimum of 1 week between) to determine the baseline concentration and week-to-week variation of the cardiac biomarkers of interest. On both trial days, different baseline characteristics will be gathered, including demographic data, clinical data, dialysis characteristics, and routine blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older.
* Clinically stable patients with end-stage renal disease treated with maintenance hemodialysis or peritoneal dialysis.
* Regarding patients treated with hemodialysis: Dialysis access with an arteriovenous fistula and able to maintain a blood flow rate >300 mL.

Exclusion Criteria:

- Not able to understand or sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Changes in the cardiac biomarkers from baseline to during and after high-flux hemodialysis and post-dilution hemodiafiltration. | Before the start of a dialysis session; after 10, 30, 60, 120, 180, and 240 minutes of dialysis; and 5-30 min. after dialysis cessation.
  Changes in the selected cardiac biomarkers from baseline, to after 10, 30, 60, 120, 180, and 240 minutes of dialysis, and 5-30 min. after dialysis cessation in both high-flux hemodialysis and post-dilution hemodiafiltration. The two dialysis modalities will be compared.

SECONDARY OUTCOMES:
Dialyzer clearance of the cardiac biomarkers in high-flux hemodialysis and post-dilution hemodiafiltration. | After 120 minutes of dialysis.
  Dialyzer clearance, calculated by dialysate and blood after 120 minutes of dialysis, of the cardiac biomarkers in high-flux hemodialysis and post-dilution hemodiafiltation. The two dialysis modalities will be compared.
Adherence of the cardiac biomarkers to the dialyzer membrane in high-flux hemodialysis and post-dilution hemodiafiltration. | After 120 minutes of dialysis.
  Adherence of the cardiac biomarkers to the dialyzer membrane after 120 minutes of dialysis in high-flux hemodialysis and post-dilution hemodiafiltation. The two dialysis modalities will be compared.

OTHER OUTCOMES:
Baseline concentrations of the cardiac biomarkers high-sensitivity cardiac troponin I, high-sensitivity cardiac troponin T, brain natriuretic peptide, and secretoneurin in patients with end-stage renal disease treated with dialysis. | Baseline.
  Concentrations of the cardiac biomarkers in patients treated with hemodialysis and peritoneal dialysis.
Week-to-week plasma variation of the cardiac biomarkers high-sensitivity cardiac troponin I, high-sensitivity cardiac troponin T, brain natriuretic peptide, and secretoneurin in patients with end-stage renal disease treated with dialysis. | At baseline on two different days with a minimum of 1 week between.
  Changes in plasma concentrations of the cardiac biomarkers at baseline on both intervention days.
Concentrations of the cardiac biomarkers high-sensitivity cardiac troponin I, high-sensitivity cardiac troponin T, brain natriuretic peptide, and secretoneurin 5-30 minutes post-dialysis. | 5-30 minutes after dialysis cessation.
  Concentrations of the cardiac biomarkers 5-30 minutes post-dialysis to investigate a potential rebound effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drivsholm CL, Nygaard L, Glerup RI, Birnum ATS, Jensen JD, Svensson M. Intradialytic kinetics of cardiac biomarkers during high-flux haemodialysis and postdilution haemodiafiltration: study protocol for a randomised crossover trial. BMJ Open. 2026 Jan 16;16(1):e105551. doi: 10.1136/bmjopen-2025-105551. PMID 41545041